CLINICAL TRIAL: NCT07310758
Title: Contrast-enhanced Ultrasound for Sentinel Node Detection in Patients With Melanoma, Breast Cancer or Head & Neck Cancer
Brief Title: Contrast-enhanced Ultrasound for Sentinel Node Detection
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N24CUS
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Breast Cancer; Head & Neck Cancer
Keywords: contrast-enhanced ultrasound
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Head and Neck Neoplasms | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-operative Sonazoid injection (Other)
  Interventions: Drug: Sonazoid

INTERVENTIONS:
Drug: Sonazoid — Intradermal injection of the ultrasound contrast agent Sonazoid.

SUMMARY:
This is a prospective single-center interventional non-inferiority study where subjects are participating for one day for patients 18 years or older with melanoma, breast cancer or head & neck cancer (including melanoma of head and neck area) and scheduled for a surgical SN procedure in the NKI-AvL without any contra-indication for Sonazoid contrast agent, such as an allergy to eggs or egg products. The primary objective is to assess the sensitivity of CEUS for intra-operative SN localization compared to the gold standard (99mTc nanocolloid). Secondary objectives are the specificity of CEUS for intra-operative SN localization, the time required to localize the SNs using CEUS and intraoperative usability of the CEUS-system. The primary endpoint is the sensitivity of the CEUS SN localization method. The conventional gamma probe will be used as ground truth comparison.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patient has been diagnosed with cancer in the skin (melanoma), breast or head & neck (including melanoma of head and neck area)
* In case of a melanoma: it should be located in the limbs or head and neck area
* Scheduled for a surgical SN procedure at the NKI-AvL
* Patient provides written informed consent

Exclusion Criteria:

* Pregnancy
* Any known clinically significant acute hypersensitivity reaction to the study medication, such as eggs or egg products
* Other contra-indications for Sonazoid contrast agent, including arteriovenous cardiac or pulmonary shunt, serious coronary arterial disease and serious pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the CEUS SN localization method | 1 day
  To assess the sensitivity of CEUS for intra-operative SN localization compared to the gold standard (99mTc nanocolloid). Could CEUS replace the conventional radioactive technetium method?

SECONDARY OUTCOMES:
Specificity of the CEUS SN localization method | 1 day
  Specificity of CEUS for intra-operative SN localization compared to the gold standard (99mTc nanocolloid)
Time in minutes | 1 day
  Time required to localize the SNs using CEUS.
System-usability score (SUS) and questionnaire for the surgeon. | 1 day
  Intraoperative usability of the CEUS-system.

CONTACTS AND LOCATIONS:
Overall Officials: Quirijn Tummers, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided